CLINICAL TRIAL: NCT02748239
Title: Evaluation of a Self-management Oriented Diabetes Education Program for the Initiation of Non-Intensive Insulin Therapy in Type 2 Diabetic Patients
Brief Title: Evaluation of a Diabetes Self-Management Education Program for Non-Intensified Insulin Therapy in Type 2 Diabetes
Acronym: MEDIAS-2-CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Forschungsinstitut der Diabetes Akademie Mergentheim (Other)
Responsible Party: Principal Investigator, Norbert Hermanns, Prof. Dr., Forschungsinstitut der Diabetes Akademie Mergentheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FIDAM-02-10
Record Dates: First submitted 2016-04-13; First posted 2016-04-22 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: diabetes self-management education; insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MEDIAS 2 CT (Active Comparator): The MEDIAS CT is a newly developed education program for the initiation of a conventional insulin therapy in type 2 diabetic patients.
  Interventions: Behavioral: MEDIAS 2 CT
- Current CT program (Placebo Comparator): This program is currently used for the initiation of conventional insulin therapy in type 2 diabetic patients.
  Interventions: Behavioral: Current CT program

INTERVENTIONS:
Behavioral: MEDIAS 2 CT — The MEDIAS 2 CT is a education program for the initiation of a conventional insulin therapy in type 2 diabetic patients. The program consists of 6 lessons and is conducted in group settings (4-8 participants).
  Arms: MEDIAS 2 CT
Behavioral: Current CT program — The Current CT program is currently used for the initiation of conventional insulin therapy in type 2 diabetic patients. The program consists of 6 lessons and is conducted in group settings (4-8 participants).
  Arms: Current CT program

SUMMARY:
A new diabetes education program for the initiation of non-intensive insulin therapy in type 2 diabetic patients (MEDIAS 2 CT) was developed.

In the evaluation, this new developed program is compared with an education programs which is currently used for diabetes education. It is expected that the new developed program (MEDIAS 2 CT) can demonstrate non-inferiority with regard to the main outcome variable glycemic control. If non-inferiority can be demonstrated superiority of this program will be tested.

DETAILED DESCRIPTION:
The MEDIAS 2 CT program is based on a self-management/empowerment approach. It is conducted as a group program comprising 6 lessons of 90 minutes each. MEDIAS 2 CT was designed to help patients perform conventional insulin therapy. In addition, MEDIAS 2 CT focused on controlling metabolic risk factors (elevated lipids and blood pressure), coping with the risk of late complications, and reducing the emotional burden of diabetes and its treatment.

The active comparator condition (ACC-CT) consisted of an established patient education program for type 2 diabetic patients with conventional insulin treatment. This education program was developed in the 1980s and 1990s and is more didactic-oriented, focusing primarily on the acquisition of knowledge, skills, and information about the correct treatment of diabetes. Both treatment arms (MEDIAS 2 CT and ACC) consisted of 6 lessons, which were conducted as group sessions.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes
* two years diabetes duration with oral treatment
* BMI > 20 and < 40 kg/m²
* written informed consent

Exclusion Criteria:

* current psychiatric disease
* dementia or other severe cognitive impairment
* severe complications
* severe conditions (e.g., cancer)
* gestational diabetes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2013-02; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
A1c values | six months follow up after termination of the programs

SECONDARY OUTCOMES:
Quality of life | six months follow up
  QoL will be assessed using the Short Form Health Survey (SF-12) questionnaire.
Diabetes knowledge | six months follow up
  A diabetes knowledge test for insulin treatment in type 2 diabetes will be used
Diabetes related emotional burden | six months follow up
  Diabetes related emotional burden / diabetes related distress will be assessed using the Problem Areas in Diabetes (PAID) questionnaire
Diabetes related distress | six months follow up
  Second questionnaire for assessing diabetes related distress is the Diabetes Distress Scale (DDS)
Self-care behavior | six months follow up
  The Summary of Diabetes Self-Care Activities (SDSCA) scale will be used.
Depression | six months follow up
  The German version of the Center of Epidemiological Studies Depression Scale (CES-D) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Hermanns, PHD, Principal Investigator — Forschungsinstitut der Diabetes Akademie Mergentheim
Locations (1):
- Diabetes Centre Mergentheim, Bad Mergentheim, Germany

IPD SHARING:
Plan to Share IPD: No